CLINICAL TRIAL: NCT07259161
Title: Prospective, Single-Arm Study on the Efficacy of a Reduced-Toxicity Conditioning Regimen Containing Thiotepa and Melphalan for Patients With Blast Phase Chronic Myeloid Leukemia
Brief Title: Modified Conditioning Regimen for CML-BP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025094
Record Dates: First submitted 2025-09-25; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: CML,Blast Phase; HSCT
MeSH Terms: interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- modified conditioning regimen (Experimental)
  Interventions: Drug: Enrolled patients with blast-phase chronic myeloid leukemia received a reduced-toxicity conditioning regimen containing thiotepa, melphalan, and fludarabine prior to undergoing allogeneic hematopoie

INTERVENTIONS:
Drug: Enrolled patients with blast-phase chronic myeloid leukemia received a reduced-toxicity conditioning regimen containing thiotepa, melphalan, and fludarabine prior to undergoing allogeneic hematopoie — This study is a prospective, interventional clinical trial recruiting patients with blast-phase chronic myeloid leukemia from the Stem Cell Transplantation Center of the Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, with an anticipated enrollment of 40 cases. Enrolled patients are scheduled to receive a reduced-toxicity conditioning regimen containing thiotepa, melphalan, and fludarabine for allogeneic hematopoietic stem cell transplantation. Thiotepa 5mg/kg on days -8 and -7, melphalan 60mg/m2 on days -5 and -4, Flu 30mg/m2 from day -6 to day -2.

SUMMARY:
Study on the Efficacy and Safety of a Reduced-Toxicity Conditioning Regimen Containing Thiotepa and Melphalan in Patients with Blast Phase Chronic Myeloid Leukemia

ELIGIBILITY:
Inclusion Criteria:

* (1) Confirmed diagnosis of blast-phase chronic myeloid leukemia, with diagnostic criteria referring to the 2020 Chinese Guidelines for Diagnosis and Treatment of Chronic Myeloid Leukemia.

Diagnostic criteria for chronic myeloid leukemia: Typical clinical manifestations combined with the presence of Philadelphia chromosome and/or BCR-ABL fusion gene positivity confirm the diagnosis.

Diagnostic criteria for blast phase:

1. Peripheral blood or bone marrow blasts ≥20%
2. Aggregates of blasts on bone marrow biopsy
3. Extramedullary blast cell infiltration (2) Age ≥18 years (3) Ability to provide self-signed informed consent (4) Must meet adequate organ function requirements:

Renal and hepatic function as follows:

AST, ALT and ALP <2× upper limit of normal (ULN) Total bilirubin <1.5× ULN Creatinine clearance >50 mL/min

Pancreatic function:

Serum amylase ≤1.5× ULN Serum lipase ≤1.5× ULN

Normal cardiac function:

Ejection fraction (EF) >60% Pulmonary artery systolic pressure ≤50 mmHg (5) HIV negative, HBV negative, HCV negative (6) Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score of 0-2 (7) Signed informed consent must be obtained before study procedures begin. For subjects aged 18 years or older, informed consent shall be signed by the patient themselves or direct family members. Considering the patient's medical condition, if the patient's own signature is medically inadvisable, the informed consent shall be signed by a legal guardian or the patient's direct family member.

Exclusion Criteria:

* 1. (1) Patients with previous autologous or allogeneic stem cell transplantation; (2) Patients concurrently diagnosed with other malignant tumors; patients assessed by investigators as having concomitant diseases that severely endanger their life safety or affect their ability to complete this study; (3) Patients with psychiatric disorders or other medical conditions that cannot comply with the requirements of study treatment and monitoring; (4) Patients unable or unwilling to sign the consent form; (5) Pregnant or lactating women; (6) Patients assessed by investigators as ineligible due to other special circumstances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2029-09-14 (Estimated); Study Completion 2029-09-14 (Estimated)

PRIMARY OUTCOMES:
overall survival, OS | 2 year

SECONDARY OUTCOMES:
Relapse free survival, RFS | 2 year
TRM | 2 year
  Treatment relater mortality
CIR | 2 year
  cumulative incidence of relapse
safety and toxicity of conditioning regimen | 2 year
  Evaluate the side effects and safety of the regimen, using Bearman score system

IPD SHARING:
Plan to Share IPD: No